CLINICAL TRIAL: NCT07224724
Title: Exosome-derived Extrahepatic Metastasis Detection By Liquid Biopsy In Colorectal Cancer Liver Metastases
Acronym: EXELION
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/EXELION
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer Liver Metastases (CRLM); Metastatic Colorectal Carcinoma (mCRC)
Keywords: CRC; Extrahepatic metastasis; liquid biopsy; Early detection
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Extrahepatic liver metastasis patients(Discovery Cohort): Patients with colorectal liver metastases (CRLM) who have confirmed extrahepatic metastasis at the time of diagnosis or treatment planning, included in the first (discovery) cohort.
- Non-extrahepatic liver metastasis patients(Discovery Cohort): Group/Cohort Description: Patients with colorectal liver metastases (CRLM) who do not have confirmed extrahepatic metastasis at the time of diagnosis or treatment planning, included in the first (discovery) cohort.
  Interventions: Other: EXELION
- Extrahepatic liver metastasis patients(Training Cohort): Extrahepatic liver metastasis patients (Training Cohort) Group/Cohort Description: Patients with colorectal liver metastases (CRLM) who have confirmed extrahepatic metastasis at the time of diagnosis or treatment planning, included in the first (training) cohort.
  Interventions: Other: EXELION
- Non-extrahepatic liver metastasis patients (Training Cohort): Group/Cohort Description: Patients with colorectal liver metastases (CRLM) who do not have confirmed extrahepatic metastasis at the time of diagnosis or treatment planning, included in the (training) cohort.
  Interventions: Other: EXELION
- Extrahepatic liver metastasis patients (Validation Cohort): Group/Cohort Description: Patients with colorectal liver metastases (CRLM) who have confirmed extrahepatic metastasis at the time of diagnosis or treatment planning, included in the second, independent, validation cohort
- Non-extrahepatic liver metastasis patients (Validation Cohort): Group/Cohort Description: Patients with colorectal liver metastases (CRLM) who do not have confirmed extrahepatic metastasis at the time of diagnosis or treatment planning, included in the second, independent, validation cohort
  Interventions: Other: EXELION

INTERVENTIONS:
Other: EXELION — A panel of exosomal microRNA, whose expression level is tested in serum or plasma
  Groups: Extrahepatic liver metastasis patients(Training Cohort); Non-extrahepatic liver metastasis patients (Training Cohort); Non-extrahepatic liver metastasis patients (Validation Cohort); Non-extrahepatic liver metastasis patients(Discovery Cohort)

SUMMARY:
Colorectal cancer is the third most common malignancy worldwide, and prognosis largely depends on how effectively metastatic disease is managed. The liver is the most frequent and prognostically important site of metastasis, and patients responding well to chemotherapy may become candidates for curative hepatic resection. However, the presence of extrahepatic metastasis (EHM) critically influences treatment eligibility and survival. Although clinical scores such as the Fong and Beppu systems include EHM as a determinant, its detection by imaging remains limited, especially for small or occult lesions. Accurate identification of EHM is also essential when considering liver transplantation for unresectable colorectal liver metastases (CRLM), where EHM remains an exclusion criterion.

The EXELION Study aims to develop a non-invasive diagnostic model using serum exosomal microRNAs (miRNAs) to detect both hepatic and extrahepatic metastases in patients with CRLM. By integrating circulating miRNA profiling with machine learning-based analysis, this study seeks to supplement imaging diagnostics, improve treatment stratification, and enhance clinical decision-making for metastatic colorectal cancer.

DETAILED DESCRIPTION:
Despite improvements in diagnostic imaging-such as CT, MRI, and PET-CT-the sensitivity of EHM detection remains limited, particularly for small or occult lesions in the lung, peritoneum, or lymph nodes. As a result, patients may be inappropriately excluded from curative surgery or exposed to non-beneficial interventions. Thus, there is a pressing need for novel, non-invasive biomarkers capable of detecting EHM with higher accuracy than imaging alone.

MicroRNAs (miRNAs), especially those encapsulated within exosomes, have emerged as stable and reproducible biomarkers reflecting tumor dynamics. Recent studies have shown that circulating miRNA signatures are associated with liver metastasis, therapeutic response, and recurrence risk in CRC. However, their utility for detecting extrahepatic metastasis has not yet been validated in clinical cohorts.

In this research effort, the investigators will leverage small RNA sequencing and machine learning to develop a predictive model for the presence of hepatic and extrahepatic metastases in patients with CRLM. The research plan will consist of three phases:

1. A discovery phase, identifying candidate miRNAs associated with the presence of EHM using next-generation sequencing (NGS) or microarray-based profiling of serum exosomal miRNAs.
2. A model development phase, establishing a quantitative reverse transcription PCR (RT-qPCR) assay and training a predictive algorithm.
3. A validation phase, independently testing the predictive accuracy of the model in an external cohort.

This diagnostic framework is provisionally termed "EXELION" (Exosome-derived Extrahepatic Metastasis Detection by LIquid Biopsy in Colorectal Cancer Liver Metastases). At the end of this study, the EXELION assay is expected to serve as a non-invasive tool to assist clinical decision-making by accurately predicting the presence of extrahepatic metastasis in patients with CRLM.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Histologically- or cytologically-confirmed colorectal cancer that is metastatic
* Availability of pre-treatment plasma samples
* Written informed consent provided
* Sufficient clinical and imaging data to determine presence/absence of extrahepatic metastasis

Exclusion Criteria:

* Prior malignancies within 5 years
* Poor sample quality or hemolysis
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with colorectal liver metastases (CRLM) originating from histologically confirmed colorectal adenocarcinoma at participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  True positive rate: the probability of a positive test result, conditioned on the individual truly being positive

SECONDARY OUTCOMES:
Specificity | Through study completion, an average of 1 year
  True negative rate: the probability of a negative test result, conditioned on the individual truly being negative
Accuracy | Through study completion, an average of 1 year
  A measure of trueness: proportion of correct predictions (both true positives and true negatives) among the total number of cases examined

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data

REFERENCES:
- [Background] Adam R, Piedvache C, Chiche L, Adam JP, Salame E, Bucur P, Cherqui D, Scatton O, Granger V, Ducreux M, Cillo U, Cauchy F, Mabrut JY, Verslype C, Coubeau L, Hardwigsen J, Boleslawski E, Muscari F, Jeddou H, Pezet D, Heyd B, Lucidi V, Geboes K, Lerut J, Majno P, Grimaldi L, Levi F, Lewin M, Gelli M; Collaborative TransMet group. Liver transplantation plus chemotherapy versus chemotherapy alone in patients with permanently unresectable colorectal liver metastases (TransMet): results from a multicentre, open-label, prospective, randomised controlled trial. Lancet. 2024 Sep 21;404(10458):1107-1118. doi: 10.1016/S0140-6736(24)01595-2. PMID 39306468
- [Background] Giuliante F, Vigano L, De Rose AM, Mirza DF, Lapointe R, Kaiser G, Barroso E, Ferrero A, Isoniemi H, Lopez-Ben S, Popescu I, Ouellet JF, Hubert C, Regimbeau JM, Lin JK, Skipenko OG, Ardito F, Adam R. Liver-First Approach for Synchronous Colorectal Metastases: Analysis of 7360 Patients from the LiverMetSurvey Registry. Ann Surg Oncol. 2021 Dec;28(13):8198-8208. doi: 10.1245/s10434-021-10220-w. Epub 2021 Jul 1. PMID 34212254
- [Background] Carpizo DR, D'Angelica M. Liver resection for metastatic colorectal cancer in the presence of extrahepatic disease. Lancet Oncol. 2009 Aug;10(8):801-9. doi: 10.1016/S1470-2045(09)70081-6. PMID 19647200
- [Background] Leung U, Gonen M, Allen PJ, Kingham TP, DeMatteo RP, Jarnagin WR, D'Angelica MI. Colorectal Cancer Liver Metastases and Concurrent Extrahepatic Disease Treated With Resection. Ann Surg. 2017 Jan;265(1):158-165. doi: 10.1097/SLA.0000000000001624. PMID 28009741
- [Background] Bojmar L, Zambirinis CP, Hernandez JM, Chakraborty J, Shaashua L, Kim J, Johnson KE, Hanna S, Askan G, Burman J, Ravichandran H, Zheng J, Jolissaint JS, Srouji R, Song Y, Choubey A, Kim HS, Cioffi M, van Beek E, Sigel C, Jessurun J, Velasco Riestra P, Blomstrand H, Jonsson C, Jonsson A, Lauritzen P, Buehring W, Ararso Y, Hernandez D, Vinagolu-Baur JP, Friedman M, Glidden C, Firmenich L, Lieberman G, Mejia DL, Nasar N, Mutvei AP, Paul DM, Bram Y, Costa-Silva B, Basturk O, Boudreau N, Zhang H, Matei IR, Hoshino A, Kelsen D, Sagi I, Scherz A, Scherz-Shouval R, Yarden Y, Oren M, Egeblad M, Lewis JS, Keshari K, Grandgenett PM, Hollingsworth MA, Rajasekhar VK, Healey JH, Bjornsson B, Simeone DM, Tuveson DA, Iacobuzio-Donahue CA, Bromberg J, Vincent CT, O'Reilly EM, DeMatteo RP, Balachandran VP, D'Angelica MI, Kingham TP, Allen PJ, Simpson AL, Elemento O, Sandstrom P, Schwartz RE, Jarnagin WR, Lyden D. Multi-parametric atlas of the pre-metastatic liver for prediction of metastatic outcome in early-stage pancreatic cancer. Nat Med. 2024 Aug;30(8):2170-2180. doi: 10.1038/s41591-024-03075-7. Epub 2024 Jun 28. PMID 38942992
- [Background] Katipally RR, Martinez CA, Pugh SA, Bridgewater JA, Primrose JN, Domingo E, Maughan TS, Talamonti MS, Posner MC, Weichselbaum RR, Pitroda SP; with the S:CORT Consortium. Integrated Clinical-Molecular Classification of Colorectal Liver Metastases: A Biomarker Analysis of the Phase 3 New EPOC Randomized Clinical Trial. JAMA Oncol. 2023 Sep 1;9(9):1245-1254. doi: 10.1001/jamaoncol.2023.2535. PMID 37471075
- [Background] Mekenkamp LJ, Haan JC, Koopman M, Vink-Borger ME, Israeli D, Teerenstra S, Ylstra B, Meijer GA, Punt CJ, Nagtegaal ID. Chromosome 20p11 gains are associated with liver-specific metastasis in patients with colorectal cancer. Gut. 2013 Jan;62(1):94-101. doi: 10.1136/gutjnl-2011-301587. Epub 2012 Jan 20. PMID 22267596
- [Background] Mahuron KM, Hernandez MC, Wong P, Fan D, Ituarte PHG, Raoof M, Singh G, Fong Y, Melstrom LG. Liver Resection With Extrahepatic Disease: A Population-Based Analysis of Thoughtful Selection. J Surg Oncol. 2025 Mar;131(3):443-449. doi: 10.1002/jso.27944. Epub 2024 Oct 28. PMID 39466980